CLINICAL TRIAL: NCT04355676
Title: A Phase 2 Randomized, Open-Label, Multicenter Study to Evaluate the Activity and Safety of Two Regimens of Low Dose Oral Selinexor in Patients With Moderate or Severe COVID-19
Brief Title: Evaluation of Activity and Safety of Two Regimens of Low Dose Oral Selinexor in Participants With Moderate or Severe COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPORT-CoV-1002
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selinexor 40mg (Experimental): Participants will receive 40 milligram (mg) of selinexor as oral tablets on Days 1 and 3 of each week for up to 2 weeks (14 days). If the participant is tolerating therapy and clinically benefitting, dosing can continue for an additional 2 weeks (28 days).
  Interventions: Drug: Selinexor
- Selinexor 20mg (Experimental): Participants will receive 20 milligram (mg) of selinexor oral tablet on Days 1, 3 and 5 of each week for up to 2 weeks (14 days). If the participant is tolerating therapy and clinically benefitting, dosing can continue for an additional 2 weeks (28 days).
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — 20 mg selinexor oral tablet.
  Other Names: KPT-330; XPOVIO

SUMMARY:
The main purpose of this study is to evaluate the activity, safety and reduction in mortality of two regimens of low dose selinexor (KPT-330) in patients with moderate or severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed laboratory diagnosis of SARS-CoV2 by standard approved reverse transcription polymerase chain reaction (RT-PCR) assay or equivalent approved testing (by local labs).
* Currently hospitalized and consented within the first 48 hours of hospitalization.
* Informed consent provided as above (patients must be dosed with study drug within 12 hours of consent).
* Has symptoms of moderate or severe COVID-19 as demonstrated by:

Moderate COVID-19:

1. Currently hospitalized and requiring medical care for COVID-19, and
2. Peripheral capillary oxygen saturation (SpO2, pulse oximetry) > 94% on room air at screening, and
3. Radiographic evidence of pulmonary infiltrates

Severe COVID-19:

1. At least one of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath at rest or with exertion, confusion, or symptoms of severe lower respiratory symptoms including dyspnea at rest or respiratory distress AND
2. Clinical signs indicative of lower respiratory infection with COVID-19, with at least one of the following: respiratory rate ≥ 30 breaths/minute (min), heart rate ≥ 125/min, Oxygen saturation (SpO2) <93% on room air or requires > 2L/minute oxygen by NC in order to maintain SaO2 ≥93%, PaO2/FiO2 <300 millimeter per mercury (mm/hg)

   * Female patients of childbearing potential must have a negative serum pregnancy test at Screening and must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.
   * Males who are sexually active must commit to use a highly effective method of contraception while receiving selinexor and for 3 months after the last selinexor dose, or consent to total sexual abstinence (abstinence must occur from enrollment and continue for 3 months after the last selinexor dose).

Exclusion Criteria:

* Evidence of critical COVID-19 based on:

  1. Respiratory failure (defined by endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula, noninvasive positive pressure ventilation, or clinical diagnosis of respiratory failure in setting of resource limitations)
  2. Septic shock (defined by SBP < 90 mm Hg, or Diastolic BP < 60 mm Hg)
  3. Multiple organ dysfunction/failure
* In the opinion of the investigator, unlikely to survive for at least 48 hours from screening or anticipate mechanical ventilation within 48 hours
* Concurrent anti-viral and/or anti-inflammatory agents (e.g., biologics, hydroxychloroquine) are not permitted.
* Inadequate hematologic parameters as indicated by the following labs:

  1. Patients with severe neutropenia (ANC <1,000 x 10^9/liter [L]) or
  2. Thrombocytopenia (e.g., platelets <100,000 per microliter of blood)
* Inadequate renal function as indicated by creatinine clearance (CrCl) <20 milliliter per minute (mL/min) using the formula of Cockcroft and Gault.
* Inadequate hepatic function defined as AST or ALT > 5x the upper limit of normal OR serum direct bilirubin > 2.5x the upper limit of normal.
* Hyponatremia defined as sodium < 135 milliequivalents per liter (mEq/L).
* In the opinion of the Investigator, patients who are below their ideal body weight and would be unduly impacted by changes in their weight.
* Unable to take oral medication when informed consent is obtained.
* Patients with a legal guardian or who are incarcerated.
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with at Least a 2 Point Improvement in the Ordinal Scale | Baseline to Day 14

SECONDARY OUTCOMES:
Time to Clinical Improvement (TTCI) | Up to Day 28
Overall Death Rate | Day 14, Day 28
Rate of Mechanical Ventilation | Up to Day 28
Time to Mechanical Ventilation | Up to Day 28
Overall Survival | Up to Day 28
Time to Improvement (2 points) in Clinical Measures Using the Ordinal Scale | Up to Day 28
Time to Intensive Care Unit (ICU) Admission | Up to Day 28
Rate of Intensive Care Unit (ICU) Admission | Up to Day 28
Length of Stay in Hospital | Up to Day 28
Percentage of Participants Discharged From Hospital | Up to Day 28
Length of Stay in Intensive Care Unit (ICU) | Up to Day 28
Duration of Oxygen Supplementation | Up to Day 28
Duration of Mechanical Ventilation | Up to Day 28
Time to Clinical Improvement in Participants ≤ 70 Years Old | Up to Day 28
Time to Clinical Improvement in Participants > 70 Years Old | Up to Day 28
Time to Clinical Improvement in Participants with Pre-existing Diseases | Up to Day 28
Change in Oxygenation Index | Up to Day 28
Time to Improvement of One Point Using WHO Ordinal Scale Improvement | Up to Day 28
Percentage of Participants Experiencing WHO Ordinal Scale Improvement of >1 point | Up to Day 28
Change from Baseline in C-reactive protein (CRP) Levels | Up to Day 28
Change from Baseline in Ferritin Levels | Up to Day 28
Change from Baseline in Lactate Dehydrogenase (LDH) Levels | Up to Day 28
Number of Participants with Adverse Events (AE) | From start of study drug administration up to follow-up (Day 30)

IPD SHARING:
Plan to Share IPD: Undecided